CLINICAL TRIAL: NCT03768609
Title: A Randomized, Open-label, Single-dose, 2-period, 2-sequence, Crossover, Phase 1 Study to Evaluate the Effect of Cyclosporine, a P-glycoprotein, Breast Cancer Resistance Protein, and Organic-anion-transporting Polypeptide Inhibitor, on the Pharmacokinetics of Pimodivir in Healthy Adult Subjects
Brief Title: A Study to Evaluate the Effect of Cyclosporine, a P-Glycoprotein, Breast Cancer Resistance Protein, and Organic-Anion-Transporting Polypeptide Inhibitor, on Pimodivir in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen-Cilag International NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CR108557; 2018-002819-10 (EudraCT Number); 63623872FLZ1015 (Other: Janssen-Cilag International NV)
Record Dates: First submitted 2018-12-06; First posted 2018-12-07 (Actual); Last update posted 2019-04-29 (Actual); Status verified 2019-04

CONDITIONS: Healthy
MeSH Terms: interventions — pimodivir; Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Sequence AB (Experimental): Participants will receive Treatment A (pimodivir 600 milligram [mg] orally as two tablets of 300 mg each) on Day 1 in Period 1 followed by Treatment B (pimodivir 600 mg as two tablets of 300 mg each plus cyclosporine 400 mg orally as four capsules of 100 mg each) on Day 1 in Period 2. Study drug intake in subsequent treatment periods will be separated by a washout period of at least 14 days.
  Interventions: Drug: Pimodivir; Drug: Cyclosporine
- Group 2: Sequence BA (Experimental): Participants will receive Treatment B on Day 1 in Period 1 followed by Treatment A on Day 1 in Period 2. Study drug intake in subsequent treatment periods will be separated by a washout period of at least 14 days.
  Interventions: Drug: Pimodivir; Drug: Cyclosporine

INTERVENTIONS:
Drug: Pimodivir — Participants will be administered pimodivir 600 mg orally as two tablets of 300 mg each.
  Other Names: JNJ-63623872
Drug: Cyclosporine — Participants will be administered cyclosporine 400 mg orally as 4 capsules of 100 mg each.
  Other Names: NEORAL

SUMMARY:
The purpose of this study is to evaluate the effect of a single oral dose of cyclosporine on the pharmacokinetics of a single oral dose of pimodivir when coadministered to healthy adult participants under fasted conditions.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to adhere to the prohibitions and restrictions specified in this protocol
* A woman of childbearing potential must have a negative highly sensitive serum (beta-human chorionic gonadotropin [beta-hCG]) at screening and on Day -1 of each treatment period
* A woman must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the study and for a period of at least 30 days after the last study drug intake
* A male participant must wear a condom when engaging in any activity that allows for passage of ejaculate to another person (male participants should also be advised of the benefit for a female partner to use a highly effective method of contraception as condom may break or leak)
* A male participant must agree not to donate sperm for the purpose of reproduction during the study and for a minimum of 90 days after last study drug intake

Exclusion Criteria:

* History of or current clinically significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders (including any abnormal bleeding or blood dyscrasias), lipid abnormalities, significant pulmonary disease, including bronchospastic respiratory disease, diabetes mellitus, hepatic or renal insufficiency (creatinine clearance below 90 milliliter per minute at screening), gastrointestinal disease (such as significant diarrhea, gastric stasis, or constipation that in the investigator's opinion could influence drug absorption or bioavailability), thyroid disease, neurologic or psychiatric disease, infection, or any other illness that the investigator considers should exclude the participant or that could interfere with the interpretation of the study results
* History of clinically significant skin disease such as, but not limited to, dermatitis, eczema, drug rash, psoriasis, food allergy, or urticaria
* Known allergies, hypersensitivity, or intolerance to pimodivir and/or cyclosporine or their excipients
* History of clinically significant drug allergy such as, but not limited to, sulfonamides and penicillins, or drug allergy diagnosed in previous studies with experimental drugs

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2018-12-06 (Actual); Primary Completion 2019-03-06 (Actual); Study Completion 2019-03-12 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | Predose, 0.5, 1, 1.5, 2, 3, 4, 5, 6 , 8, 12, 16, 24, 48, 72, 96, 120, 144, 168 hours postdose on Day 8
  Cmax is defined as maximum observed plasma concentration.
Area Under the Plasma Concentration-Time Curve From Time Zero to Last Quantifiable Concentration Time (AUC [0-Last]) | Predose, 0.5, 1, 1.5, 2, 3, 4, 5, 6 , 8, 12, 16, 24, 48, 72, 96, 120, 144, 168 hours postdose on Day 8
  AUC(0-Last) is area under the plasma concentration-time curve from time zero to time of the last measurable (non-below quantification limit) concentration, calculated by linear-linear trapezoidal summation.
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC [0-infinity]) | Predose, 0.5, 1, 1.5, 2, 3, 4, 5, 6 , 8, 12, 16, 24, 48, 72, 96, 120, 144, 168 hours postdose on Day 8
  AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC(last) and C(last)/lambda(z); where C(last) is the last observed measurable (non-below quantification limit) concentration.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events (AEs) as a Measure of Safety and Tolerability | Approximately 65 days
  An AE is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non investigational) product. An AE does not necessarily have a causal relationship with the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag International NV Clinical Trial, Study Director — Janssen-Cilag International NV
Locations (1):
- Clinical Pharmacology Unit, Merksem, Belgium

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials\transparency. As noted on this site, requests for access to the study data can be submitted through Yale open Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency